CLINICAL TRIAL: NCT07193888
Title: Navitor Japan Post-Market Study
Brief Title: Navitor Japan Study
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10599
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Severe Aortic Stenosis
Keywords: NAVITOR; Transcatheter aortic valve implantation (TAVI); Aortic Stenosis; Cardiovascular Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Cohort 1: This study will enroll subjects of all genders from the population of patients qualifying for TAVI.
  Interventions: Device: Navitor Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Device: Navitor Transcatheter Aortic Valve Implantation — Subjects will undergo transcatheter aortic valve implantation (TAVI) with the Navitor valve, the FlexNav Delivery system and the Navitor Loading System.
  Other Names: TAVI

SUMMARY:
The Navitor Japan Study is designed to evaluate the safety and performance of the Navitor™ valve used in combination with the FlexNav™ delivery system in a contemporary, real-world setting.

DETAILED DESCRIPTION:
A prospective, single-arm, observational, multicenter post-market clinical study enrolling approximately 100 Japanese patients with symptomatic, severe aortic stenosis. The study will evaluate the safety and performance of the Navitor TAVI system, including future commercially available iterations, as they become available in Japan. Enrolled subjects will undergo follow-up at discharge, 30 days and 1-year post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eligible per the current approved indication after Heart Team discussion and intended to undergo a Navitor TAVI procedure.
2. The patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent as approved by the EC of the respective clinical site.
3. The patient and the treating physician agree that the subject will return for all required post-procedure follow-up visits

Exclusion Criteria:

1. Patient is not eligible for the Navitor TAVI System per the current Instructions for Use (IFU).
2. Life expectancy < 12 months from the time of informed consent due to non-cardiac co-morbid conditions.
3. In the judgment of the Investigator, patient presents with a medical, social, or psychological condition that could limit the ability or willingness to participate in the study, comply with study required testing and/or follow-up visits or that could impact scientific integrity of the study.
4. Known contraindication for computed tomography (CT) or sensitivity to contrast media, which cannot be adequately premedicated.
5. Inability to tolerate antiplatelet/anticoagulation therapy or nitinol alloy (nickel and titanium), which cannot be adequately premedicated.
6. Currently participating in an investigational drug or device study that may confound the results of this study.
7. Anatomy that makes insertion and endovascular access to the aortic valve difficult and/or impossible.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic, severe aortic stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 30 days post index procedure
  The primary safety endpoint is all-cause mortality at 30 days post-TAVI procedure, which will be assessed descriptively
Primary Performance Endpoint | 30 days post index procedure
  The primary performance endpoint is moderate or greater paravalvular leak (PVL) at 30 days as measured on a transthoracic echocardiogram (TTE) by the echocardiographic core laboratory. This endpoint will be reported as % subjects with moderate or greater PVL at 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka Keisatsu Hospital, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No